CLINICAL TRIAL: NCT03392662
Title: Hemopatch Performance Evaluation: A Prospective Observational Registry
Status: Completed | Type: Observational
Sponsor: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: BXU011443
Record Dates: First submitted 2017-12-19; First posted 2018-01-08 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Dura Mater Nick Cut or Tear; Hemostatis; Air Leakage; Body Fluid Leakage
MeSH Terms: conditions — Lacerations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (6):
- Hemopatch Sealant Use with Hepatobiliary Surgery
  Interventions: Device: Hemopatch
- Hemopatch Sealant Use with General Surgery
  Interventions: Device: Hemopatch
- Hemopatch Sealant Use with Lung Surgery
  Interventions: Device: Hemopatch
- Hemopatch Sealant Use with Cardiovascular Surgery
  Interventions: Device: Hemopatch
- Hemopatch Sealant Use with Neurological/Spinal Surgery
  Interventions: Device: Hemopatch
- Hemopatch Sealant Use with Urologic Surgery
  Interventions: Device: Hemopatch

INTERVENTIONS:
Device: Hemopatch — Patients received product at the discretion of their surgeon.

SUMMARY:
To assess the clinical performance and safety of HEMOPATCH Sealing Hemostat in a post-marketing setting in cardiovascular, thoracic, urologic, neurological, and other general surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients of any age
* Patients who had undergone open or minimal invasive surgical (MIS) procedures requiring the use of a patch to achieve dura repair, hemostasis, or control of leakage of air or other body fluid when pressure, ligature or other conventional procedures had been ineffective or impractical and where use of hemopatch was deemed appropriate by the surgeon according to its IFU in the following organ systems:

  1. Hepato-biliary (liver, pancreas, gallbladder)
  2. General surgery (in thyroid and other regions)
  3. Cardiovascular (heart and vessels)
  4. thoracic (lung and mediastinum)
  5. Urological (kidney, prostate, and bladder
  6. Neurological (dura mater, brain and spinal cord)
* Provision of written informed consent/assent, as applicable, up to 72 hours after the date of surgery

Exclusion Criteria:

* Patients with known hypersensitivity to bovine proteins or brilliant blue
* Patients who had intraoperative pulsatile or severe bleeding at the target application site (TAS)
* Patients who had an active infection at the TAS

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient who had undergone a general, cardiovascular, thoracic, urological, or neurological surgery during which the use of a patch was required to repair the dura or to achieve hemostasis, control leakage of air or other body fluid because pressure, ligature or conventional procedures were ineffective or impractical and during which Hemopatch was used according to Instructions for use.
Sampling Method: Probability Sample
Enrollment: 621 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2019-01-28 (Actual); Study Completion 2019-01-28 (Actual)

PRIMARY OUTCOMES:
Percentage of patients achieving hemostasis after 2 minutes of surgery | Day 1 (up to 2 minutes postoperative)
Percentage of patients achieving hemostasis without re-bleeding at the time of surgical closure | Day 1 (intraoperative)
Absence of air leak in lung at time of surgical closure | Day 1 (intraoperative)
Tight closure achieved in dura mater at time of surgical closure | Day 1 (intraoperative)
  No leak after inspection per local standard of care
Number of patients with chest tube drainage >=5 days after thoracic/lung surgery | Day 5 up to 4 weeks (postoperative)
Number of patients needing reinsertion of chest tube for pneumothorax after thoracic/lung surgery | Up to 4 weeks (postoperative)
Number of patients with postoperative pancreatic fistulas after hepatobiliary surgery | Up to 4 weeks (postoperative)
Duration of bile leakage after hepatobiliary surgery | Up to 4 weeks (postoperative)
Number of patients with postoperative cerebrospinal fluid (CSF) leakage after neurological surgery | Up to 4 weeks (postoperative)
  External or internal accumulation including pseudomeningocele
Number of patients with postoperative urinary fistula formation after urological surgery | Up to 4 weeks (postoperative)
Gastrointestinal anastomosis leakage/fistula after general surgery | Up to 4 weeks (postoperative)
Number of patients with related Adverse Events | Up to 4 weeks (postoperative)

SECONDARY OUTCOMES:
Number of Hemopatch units applied | Up to 4 weeks (postoperative)
Surgical revisions/reoperations due to bleeding, air, or other body fluid leakage | Up to 4 weeks (postoperative)
Number of intraoperative transfusions by type and amount of blood product transfused | Day 1 (intraoperative)
  Unit of measure will be number of transfusion procedures and will be summarized as a single outcome measure.
Number of postoperative transfusions by type and amount of blood product transfused up to 72 hours after surgery | Up to 72 hours (postoperative)
  Unit of measure will be number of transfusion procedures and will be summarized as a single outcome measure.
Surgery duration | Day 1 (intraoperative)
Length of hospital stay | Up to 4 weeks (postoperative)
  Intensive Care Unit (ICU) and hospital
Ease of product preparation | Day 1 (intraoperative)
  Surgeon's overall product assessment and satisfaction recorded on questionnaire.
Ease of product handling | Day 1 (intraoperative)
  Surgeon's overall product assessment and satisfaction recorded on questionnaire.
Assessment of product tissue adherence | Day 1 (intraoperative)
  Surgeon's overall product assessment and satisfaction recorded on questionnaire.
Surgeon's overall satisfaction of product | Day 1 (intraoperative)
  Surgeon's overall product assessment and satisfaction recorded on questionnaire.
Product characteristics appreciated by Surgeon | Day 1 (intraoperative)
  Surgeon's overall product assessment and satisfaction recorded on questionnaire.
Product characteristics liked least by Surgeon | Day 1 (intraoperative)
  Surgeon's overall product assessment and satisfaction recorded on questionnaire.

CONTACTS AND LOCATIONS:
Locations (15):
- Innsbruck Universitaetsklinik, Innsbruck, Austria
- Czechia (4):
  - Fakultní nemocnice u sv. Anny v Brně, Brno
  - Krajská Nemocnice Liberec, Liberec
  - Fakultní Nemocnice Ostrava, Ostrava
  - Thomayerova Nemocnice, Prague
- Germany (4):
  - Marien-Krankenhaus Bergisch Gladbach, Bergisch Gladbach
  - Deutsches Herzzentrum Berlin, Berlin
  - ASKLEPIOS Klinik St. Georg, Hamburg
  - Universitaetsklinikum Regensburg, Regensburg
- Azienda Ospedaliero-Universitaria Careggi, Florence, Italy
- Spain (5):
  - Hospital de Vall d'Hebrón, Barcelona
  - Hospital Universitari de Girona Doctor Josep Trueta, Girona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital La Paz, Madrid
  - Hospital Universitario Virgen del Rocio, Seville

REFERENCES:
- [Background] Lombardo C, Lopez-Ben S, Boggi U, Gutowski P, Hrbac T, Krska L, Marquez-Rivas J, Russello D, York E, Zacharias M. Hemopatch(R) is effective and safe to use: real-world data from a prospective European registry study. Updates Surg. 2022 Oct;74(5):1521-1531. doi: 10.1007/s13304-022-01353-y. Epub 2022 Aug 20. PMID 35986865